CLINICAL TRIAL: NCT07223736
Title: Postpartum Education Via Artificial Intelligence for Recovery and Loneliness (PEARL): A Randomized Controlled Trial
Brief Title: Postpartum Education Via Artificial Intelligence for Recovery and Loneliness: A Randomized Controlled Trial
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cecile Ferrando, Professor OBGYN & Reproductive Sciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 812859
Record Dates: First submitted 2025-10-31; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pelvic Floor Disorder; Loneliness; Postpartum; Mental Health; Depression; Peritraumatic Distress; Women; Artificial Intelligence (AI); Chatbot
Keywords: loneliness; postpartum; pelvic floor disorder; mental health; depression; peritraumatic distress; artificial intelligence; AI; chatbot; LLM; women; large language model
MeSH Terms: conditions — Pelvic Floor Disorders; Psychological Well-Being; Depression | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either standard postpartum care alone or the chatbot intervention in addition to standard postpartum care. The intervention group will have access to the chatbot for a 4-week period. No crossover between groups will occur. Outcomes will be assessed at baseline, post-intervention, and at 6 months postpartum for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard postpartum care (Active Comparator): Standard postpartum care
  Interventions: Other: Standard of Care (SOC)
- Generative AI Chatbot Intervention (Experimental): Generative AI Chatbot Intervention
  Interventions: Other: Generative artificial intelligence (genAI) postpartum chatbot; Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Generative artificial intelligence (genAI) postpartum chatbot — Participants randomly assigned to the chatbot intervention will be provided a URL to a secure, HIPAA-compliant web application hosted by UC San Diego (https://knolohealth.org/). This application features a generative AI-powered chatbot designed to deliver postpartum pelvic floor education and support. The chatbot is available for a 4-week period following enrollment and can be accessed at any time during that window.
  The chatbot's educational content is grounded in reputable, evidence-based resources, including national and international urogynecology patient education materials, as well as postpartum recovery guidelines. Participants can interact with the chatbot to ask questions and will receive tailored educational responses related to pelvic floor health.
  No additional in-person study visits are required for the intervention. Chatbot usage data (e.g., frequency, timing and content of chatbot interactions) will be collected to assess engagement and user needs.
  Arms: Generative AI Chatbot Intervention
Other: Standard of Care (SOC) — Access to the same postpartum care that participants would receive if they did not participate in the study.
  Other Names: Standard postpartum care; Routine postpartum care

SUMMARY:
The goal of this clinical trial is to learn whether a postpartum chatbot powered by generative artificial intelligence (genAI) can help new mothers get better pelvic floor health information and feel less lonely after childbirth.

The main questions this study aims to answer are:

* Does using the chatbot improve postpartum pelvic floor health knowledge?
* Does using the chatbot help reduce feelings of loneliness during the postpartum period?
* Does using the chatbot impact pelvic floor symptoms?

Researchers will compare standard postpartum care to standard care plus the chatbot.

Participants will:

Be assigned by chance (like flipping a coin) to standard postpartum care with or without access to the chatbot.

If in the chatbot group, participants will receive education and support via the chatbot over a 4-week period.

Both groups will complete questionnaires to measure their pelvic floor knowledge, pelvic floor symptoms, feelings of loneliness, depression, infant bonding, perceived social support, adverse childhood experiences, and peri-traumatic distress.

The chatbot was created by urogynecology experts in collaboration with UC San Diego computer science and biomedical informatics researchers. The chatbot is designed to give new mothers personalized, evidence-based information and support in real time.

DETAILED DESCRIPTION:
Pelvic floor disorders (PFDs)-including urinary incontinence, fecal incontinence, and pelvic organ prolapse-are highly prevalent and debilitating conditions affecting approximately 25% of women in the United States.Pregnancy and childbirth are known risk factors for developing PFDs. Recent imaging studies show that injuries to the levator ani muscle, perineal body, and perineal membrane occur in up to 19% of first-time mothers. Urogynecologic conditions, such as urinary and bowel incontinence, are common after pregnancy and often result in a catastrophic impact on maternal quality of life not just because of the physical symptoms, but also because of the associated embarrassment, isolation, and negative stigma.Compounding this challenging recovery further, one in five women will experience a perinatal mood disorder, such as anxiety, depression, or PTSD. Despite the profound physical and psychological impacts of childbirth, postpartum care remains limited, inconsistent, and difficult to access.

It is well established that many postpartum individuals seek education, community, and emotional validation on various online platforms. When postpartum individuals are interviewed, many report feeling their postpartum health concerns are neglected and minimized, resulting in feelings of disempowerment through the help-seeking process. Further compounding these feelings, is the lack of timely or frequent postpartum care with many women having difficulty attending postpartum visits and often being only seen once postpartum. Furthermore, patients who experience a severe pelvic floor injury at delivery may not have access to specialty care clinic for peripartum pelvic floor disorders. Through qualitative interviews with postpartum individuals with obstetric anal sphincter injury (OASI), themes of seeking social support through online communities such as Facebook and Instagram were identified, though the effectiveness of these groups in meeting patients' needs is unclear. While social media platforms may serve as a support bridge for patients as they await their postpartum visit, much of the content on these platforms is anecdotal, humorous, and not produced by physicians. Furthermore, these platforms also expose recovering individuals to distressing anecdotal narratives or idyllic imagery that may further worsen mental health in this vulnerable patient population.

As postpartum individuals navigate the fourth trimester, feelings of loneliness and isolation are common. Loneliness is linked to adverse health outcomes, including cardiovascular disease, cognitive health, infectious disease, and all-cause mortality, yet its impact on pelvic floor muscle recovery remains largely unexplored.In the U.S. Surgeon General's 2023 advisory, the healing power of social connection and community was emphasized. Lunstad et al., acknowledge that despite mounting evidence healthcare has been slow to recognize that social relationships are health determinants. Postpartum individuals are not immune to loneliness, in fact in a systematic review, the prevalence of loneliness among peripartum women ranged between 32% to 100%. Identifying solutions to address the epidemic of postpartum loneliness is critical to improving the overall health of both birthing individuals and their infants.

Optimizing postpartum maternal mental and physical health is not only critical for the postpartum individual's recovery, but also profoundly influences infant development. The first weeks and months after delivery represent a sensitive window for neonatal brain development, attachment formation, and physiological regulation. When postpartum individuals experience persistent pain, incontinence, or limited mobility, it can hinder early caregiving, reduce breastfeeding success, and increase maternal-infant separation.Maternal mental health disorders have been associated with disrupted bonding, impaired infant stress regulation, and long-term cognitive, emotional, and behavioral challenges in children. Emerging research in developmental neuroscience demonstrates that early maternal-infant interactions shape the infant's stress response system and neurodevelopment trajectory through mechanisms involving cortisol regulation, oxytocin signaling, and epigenetic modifications. It is possible that through improved maternal knowledge of pelvic floor health, that postpartum individuals will experience improved self-efficacy, decreased loneliness, and possibly even improved physical recovery.

However, peripartum pelvic floor disorder knowledge is lacking. McLennan et al., evaluated the information that patients received during pregnancy, and found that the most neglected content area was education on PFDs. Furthermore, Reagan et al., found that most available patient education materials are above the reading level recommended by the National Institutes of Health for maximum patient comprehension. Numerous publications have concurred that there is a global lack of knowledge and understanding of urinary incontinence, pelvic organ prolapse, and bowel incontinence educating patients on PFDs, with many authors calling for increased emphasis of pelvic floor health and development of educational programs to inform patients.Rutledge et al., performed a randomized controlled trial assessing peripartum pelvic floor health knowledge as measured with the Prolapse and Incontinence Knowledge Questionnaire (PIKQ) among women randomized to receiving written handouts only or written handouts plus an interactive workshop. Results of this study demonstrated that both groups improved in their knowledge, but interestingly patient perspectives on preferred education was discovered. Themes surrounding the delivery of educational content were identified, such as a preference for reviewing informational materials on their own time and having the opportunity to receive real-time responses to questions. In addition, themes of preferred educational content developed, including desire to understand the etiology of PFDs, comfort with discussing PFDs, and relief in learning treatment options.

While in person support groups, text based platforms, and telehealth coaches have attempted to address this unmet need for postpartum support and education, conversational agents (chatbots) have recently emerged as a promising tool for scalable, real-time health education and support in this patient population. Chatbots have the potential to deliver just-in-time adaptive intervention (JITAI), a novel intervention design that adapts the provision of support (ie type, timing, intensity) to delivery support at the moment and in the context that the user needs it most. JITAI increases user receptivity to support and is increasingly being used to help support health behavior changes, including mental health. Using natural language processing, chatbots interact with users to provide education, emotional support, and symptom guidance. Their availability on smartphones has made them a widely used tool for health information retrieval and mental wellness. Prior studies evaluating chatbots in the peripartum period have demonstrated successful engagement of individuals, improved user knowledge, and reduction in depressive symptoms. Furthermore, outside of the peripartum patient population, chatbots are known to reduce loneliness through direct companionship and social interactions. Kim et al., explored the mental health potential of AI social chatbots over four weeks and found that UCLA loneliness scores started to improve by week two among individuals interacting with the chatbot. Thus, we propose a similar study intervention time frame (4 weeks).

There is an urgent, unmet need for comprehensive, real time postpartum pelvic floor health education and support in the immediate postpartum period. To address this unmet need, we have developed a genAI postpartum chatbot to bridge the gap for patients to their providers. The chatbot was built using UCSD Health approved Large Language Models (LLMs) made available within the UCSD Health Cloud. In order to provide accurate curated information in response to patient questions in the chatbot, the chatbot implements retrieval augmented generation (RAG).

In the setting of rising maternal morbidity, coupled with limited healthcare access, understanding the impact of a postpartum educated AI chatbot on maternal loneliness, knowledge, and physical recovery is critical to improve maternal and infant health.

ELIGIBILITY:
Inclusion Criteria:

1. Has the capacity to provide informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Postpartum persons, aged >18 years old
4. Primiparous
5. Vaginal or cesarean delivery
6. English Speaking
7. Internet access and proficiency of internet access
8. Access to a smartphone
9. Postpartum 2-6 weeks

Exclusion Criteria:

1. Multiparous
2. Major neonatal anomaly
3. Delivery < 34 weeks gestational age
4. Intrauterine fetal demise (IUFD)
5. Enrollment in any interfering studies
6. Unanticipated NICU admission
7. Discharge home without live baby
8. Surrogates/gestational carrier
9. Birthing individuals with baby placed for adoption
10. Currently pregnant
11. Psychiatric history requiring psychiatric hospitalization prior to delivery
12. Other psychiatric conditions needing immediate attention and intervention as determined by study team and/or treatment team

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Prolapse and incontinence knowledge | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  Prolapse and incontinence knowledge will be assessed via the validated prolapse and incontinence knowledge questionnaire (PIKQ). This is a validated, self-administered instrument designed to assess women's knowledge about the epidemiology, pathogenesis, diagnosis, and treatment of pelvic organ prolapse and urinary incontinence. The PIKQ has been used in the postpartum population.This questionnaire consists of two 12 item sub-scales (total of 24 questions) with answer options of "agree", "disagree", or "don't know". Correct answers receive 1 point, while incorrect answers receive 0 points. Sub-scale score ranges from 0-12 and total score ranges from 0-24. Higher scores indicate more knowledge. We aim to detect a clinically meaningful difference of 4 points between the control and intervention group. This 4-point difference represents approximately a 17% increase in knowledge and is considered a reasonable effect based on prior literature and the nature of the educational intervention.

SECONDARY OUTCOMES:
Loneliness scores | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  Loneliness will be assessed via the revised UCLA loneliness scale. The revised UCLA loneliness scale provides a robust, sensitive measure of loneliness with high internal consistency and validity, and has been used in the postpartum population.This 20 question scale measures subjective feelings of loneliness and social isolation. Responses are rated on a 4 point scale; "1=never", "2=rarely", "3=sometimes", "4=often" with total score ranges from 20 to 80. Higher scores indicate worse loneliness.
Pelvic Floor Distress | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  Pelvic floor distress will be assessed via the Pelvic Floor Distress Inventory-20 (PFDI-20). This is a validated questionnaire that assesses the presence and impact of PFD symptoms in women. It is divided into 3 validated sub-scales to assess pelvic organ prolapse distress (POPDI-6), colorectal-anal distress (CRADI-8), and urinary distress (UDI-6). Each item is scored from 0 (not at all) to 4 (quite a bit) and the mean of each sub-scale is multiplied by 25 to obtain a sub-scale range from 0 to 100 and a total PFD-20 scores of 0 to 300.

OTHER OUTCOMES:
Patient global impression of improvement (PGI-I) | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  PGI-I asks patients to rate their overall improvement after an intervention compared to their baseline state, using a 7-point Likert scale from "very much better" to "very much worse." It is designed to capture the patient's perception of change specifically attributable to an intervention, making it highly relevant for assessing treatment outcomes in urogynecology.
Mother to Infant Bonding Scale (MIBS) | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  The Mother to Infant Bonding Scale (MIBS) is 8 question scale designed to measure maternal emotion towards their infant. Each item is scores on a 4-point Likert scale (0 = Not at all, 1 = A little, 2 = Quite a lot, 3 = Very much). Scores range 0 to 24, with higher scores indicating greater difficulties in mother-infant bonding.
Peritraumatic Distress Inventory (PDI) | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  The Peritraumatic Distress Inventory (PDI) is a validated, self-report questionnaire designed to assess emotional and physiological distress experienced during or immediately after a traumatic event. This 13-item self-report questionnaire uses a 5-point Likert scale (0 = Not at All True, 1 = Slightly True, 2 = Somewhat True, 3 = Very True, and 4 = Extremely True to assess responses). The items are summed to achieve total scores in the range 0 to 52. The PDI has been evaluated in the postpartum setting and a score of 15+ on the modified PDI (exclusion of item 4 "I felt afraid for my own safety") produced high sensitivity and specificity: 88% with a positive CB-PTSD screen in the first postpartum months and 93% with a negative screen.
Edinburgh Postnatal Depression Scale (EPDS) | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  The Edinburgh Postnatal Depression Scale (EPDS) screens for symptoms of postpartum depression and anxiety over the past 2 weeks and has a score range of 0 to 30, with a score of > 10 indicating possible depression. It is a validated survey in antenatal populations as well.
Multidimensional Scale of Perceived Social Support (MSPSS) | Will be administered to both groups at three time points: 1) at enrollment, 2) post-intervention or standard of care, 3) at 6 months postpartum.
  The Multidimensional Scale of Perceived Social Support (MSPSS) is 12 item scale on perception of perceived adequacy of social support from friends, family and significant other. There are 4 items per sub-scale and items are scores on a 7-point Likert Scale (1 = very strongly disagree to 7 = very strongly agree). Higher scores indicate greater perceived social support.
Adverse Childhood Experience (ACE) Questionnaire | Will be administered to both groups at a single time point: at enrollment.
  The Adverse Childhood Experience (ACE) Questionnaire consists of 10 items covering three domains: abuse (emotional, physical, sexual), neglect (emotional, physical), and household challenges (parental separation/divorce, domestic violence, substance abuse, mental illness, incarceration). Respondents answer yes/no to each item, and the total ACE score reflects the number of categories experienced. Higher scores are associated with increased risk for a range of adverse health outcomes in adulthood, including mental illness, substance use, and chronic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Single site location and current IRB approval is for no data sharing.

REFERENCES:
- [Background] Can FG, Akis G, Solmaz E. The effect of the level of perceived social support in the postpartum period on maternal functioning and maternal attachment. J Pediatr Nurs. 2024 Nov-Dec;79:e192-e202. doi: 10.1016/j.pedn.2024.10.021. Epub 2024 Oct 29. PMID 39472191
- [Background] Canty-Mitchell J, Zimet GD. Psychometric properties of the Multidimensional Scale of Perceived Social Support in urban adolescents. Am J Community Psychol. 2000 Jun;28(3):391-400. doi: 10.1023/A:1005109522457. PMID 10945123
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Jagodnik KM, Ein-Dor T, Chan SJ, Titelman Ashkenazy A, Bartal A, Barry RL, Dekel S. Screening for post-traumatic stress disorder following childbirth using the Peritraumatic Distress Inventory. J Affect Disord. 2024 Mar 1;348:17-25. doi: 10.1016/j.jad.2023.12.010. Epub 2023 Dec 7. PMID 38070747
- [Background] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Background] Chiu JL, Wei LC. Loneliness as a Predictor of Disability in Older Adults: Implications of the UCLA Loneliness Scale Cutoff Score Across Cultural Contexts. Int J Geriatr Psychiatry. 2024 Nov;39(11):e70011. doi: 10.1002/gps.70011. PMID 39516187
- [Background] Gosling CJ, Colle R, Cartigny A, Jollant F, Corruble E, Frajerman A. Measuring loneliness: a head-to-head psychometric comparison of the 3- and 20-item UCLA Loneliness Scales. Psychol Med. 2024 Oct 31;54(14):1-7. doi: 10.1017/S0033291724002083. Online ahead of print. PMID 39479755
- [Background] Shah AD, Massagli MP, Kohli N, Rajan SS, Braaten KP, Hoyte L. A reliable, valid instrument to assess patient knowledge about urinary incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1283-9. doi: 10.1007/s00192-008-0631-x. Epub 2008 May 15. PMID 18480958
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Suharwardy S, Ramachandran M, Leonard SA, Gunaseelan A, Lyell DJ, Darcy A, Robinson A, Judy A. Feasibility and impact of a mental health chatbot on postpartum mental health: a randomized controlled trial. AJOG Glob Rep. 2023 Mar 29;3(3):100165. doi: 10.1016/j.xagr.2023.100165. eCollection 2023 Aug. PMID 37560011
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Kim M, Lee S, Kim S, Heo JI, Lee S, Shin YB, Cho CH, Jung D. Therapeutic Potential of Social Chatbots in Alleviating Loneliness and Social Anxiety: Quasi-Experimental Mixed Methods Study. J Med Internet Res. 2025 Jan 14;27:e65589. doi: 10.2196/65589. PMID 39808786
- [Background] Gasteiger N, Loveys K, Law M, Broadbent E. Friends from the Future: A Scoping Review of Research into Robots and Computer Agents to Combat Loneliness in Older People. Clin Interv Aging. 2021 May 24;16:941-971. doi: 10.2147/CIA.S282709. eCollection 2021. PMID 34079242
- [Background] Laranjo L, Dunn AG, Tong HL, Kocaballi AB, Chen J, Bashir R, Surian D, Gallego B, Magrabi F, Lau AYS, Coiera E. Conversational agents in healthcare: a systematic review. J Am Med Inform Assoc. 2018 Sep 1;25(9):1248-1258. doi: 10.1093/jamia/ocy072. PMID 30010941
- [Background] McAlister K, Baez L, Huberty J, Kerppola M. Chatbot to Support the Mental Health Needs of Pregnant and Postpartum Women (Moment for Parents): Design and Pilot Study. JMIR Form Res. 2025 Apr 8;9:e72469. doi: 10.2196/72469. PMID 40202166
- [Background] Ben-Zeev D, Kaiser SM, Brenner CJ, Begale M, Duffecy J, Mohr DC. Development and usability testing of FOCUS: a smartphone system for self-management of schizophrenia. Psychiatr Rehabil J. 2013 Dec;36(4):289-296. doi: 10.1037/prj0000019. Epub 2013 Sep 9. PMID 24015913
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Amil S, Da SM, Plaisimond J, Roch G, Sasseville M, Bergeron F, Gagnon MP. Interactive Conversational Agents for Perinatal Health: A Mixed Methods Systematic Review. Healthcare (Basel). 2025 Feb 8;13(4):363. doi: 10.3390/healthcare13040363. PMID 39997238
- [Background] Inkster B, Kadaba M, Subramanian V. Understanding the impact of an AI-enabled conversational agent mobile app on users' mental health and wellbeing with a self-reported maternal event: a mixed method real-world data mHealth study. Front Glob Womens Health. 2023 Jun 2;4:1084302. doi: 10.3389/fgwh.2023.1084302. eCollection 2023. PMID 37332481
- [Background] Teoule J, Woll C, Ray J, Sutterlin M, Filsinger B. The effectiveness of integrated online health-coaching on physical activity and excessive gestational weight gain: a prospective randomized-controlled trial. Arch Gynecol Obstet. 2024 Jul;310(1):307-314. doi: 10.1007/s00404-023-07296-y. Epub 2024 Jan 13. PMID 38217763
- [Background] Bravata DM, Kim J, Russell DW, Goldman R, Pace E. Digitally Enabled Peer Support Intervention to Address Loneliness and Mental Health: Prospective Cohort Analysis. JMIR Form Res. 2023 Nov 6;7:e48864. doi: 10.2196/48864. PMID 37930770
- [Background] Uscher-Pines L, Kapinos K, Waymouth M, Howell K, Alvarado G, Ray K, Demirci J, Mehrotra A, Rogers R, James KF, DeYoreo M. Telelactation Services and Breastfeeding by Race and Ethnicity: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2461958. doi: 10.1001/jamanetworkopen.2024.61958. PMID 40014345
- [Background] Chae SY, Chae MH, Kandula S, Winter RO. Promoting improved social support and quality of life with the CenteringPregnancy(R) group model of prenatal care. Arch Womens Ment Health. 2017 Feb;20(1):209-220. doi: 10.1007/s00737-016-0698-1. Epub 2016 Dec 17. PMID 27988822
- [Background] Rutledge E, Spiers A, Vardeman J, Griffin N, Nisar T, Muir T, Antosh DD. Educating Women About Pelvic Floor Disorders During Pregnancy From the First to the "Fourth Trimester": A Randomized Clinical Trial. Urogynecology (Phila). 2023 Sep 1;29(9):770-776. doi: 10.1097/SPV.0000000000001341. PMID 37607311
- [Background] Toprak Celenay S, Coban O, Korkut Z, Alkan A. Do community-dwelling pregnant women know about pelvic floor disorder? Women Health. 2021 Jul;61(6):609-616. doi: 10.1080/03630242.2021.1942398. Epub 2021 Jun 17. PMID 34139962
- [Background] Liu J, Tan SQ, Han HC. Knowledge of pelvic floor disorder in pregnancy. Int Urogynecol J. 2019 Jun;30(6):991-1001. doi: 10.1007/s00192-019-03891-3. Epub 2019 Feb 19. PMID 30783706
- [Background] Mandimika CL, Murk W, Muhlhauser McPencow A, Lake A, Wedderburn T, Collier CH, Connell KA, Guess MK. Knowledge of pelvic floor disorders in a population of community-dwelling women. Am J Obstet Gynecol. 2014 Feb;210(2):165.e1-9. doi: 10.1016/j.ajog.2013.10.011. Epub 2013 Oct 11. PMID 24126299
- [Background] Reagan KM, O'Sullivan DM, Harvey DP, Lasala CA. Readability of patient information pamphlets in urogynecology. Female Pelvic Med Reconstr Surg. 2015 Mar-Apr;21(2):63-5. doi: 10.1097/SPV.0000000000000152. PMID 25679357
- [Background] McLennan MT, Melick CF, Alten B, Young J, Hoehn MR. Patients' knowledge of potential pelvic floor changes associated with pregnancy and delivery. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jan;17(1):22-6. doi: 10.1007/s00192-005-1325-2. Epub 2005 Jul 8. PMID 16003482
- [Background] Essex MJ, Boyce WT, Hertzman C, Lam LL, Armstrong JM, Neumann SM, Kobor MS. Epigenetic vestiges of early developmental adversity: childhood stress exposure and DNA methylation in adolescence. Child Dev. 2013 Jan-Feb;84(1):58-75. doi: 10.1111/j.1467-8624.2011.01641.x. Epub 2011 Sep 2. PMID 21883162
- [Background] Champagne FA. Epigenetic influence of social experiences across the lifespan. Dev Psychobiol. 2010 May;52(4):299-311. doi: 10.1002/dev.20436. PMID 20175106
- [Background] Rogers AM, Youssef GJ, Teague S, Sunderland M, Le Bas G, Macdonald JA, Mattick RP, Allsop S, Elliott EJ, Olsson CA, Hutchinson D. Association of maternal and paternal perinatal depression and anxiety with infant development: A longitudinal study. J Affect Disord. 2023 Oct 1;338:278-288. doi: 10.1016/j.jad.2023.06.020. Epub 2023 Jun 9. PMID 37302506
- [Background] Slomian J, Honvo G, Emonts P, Reginster JY, Bruyere O. Consequences of maternal postpartum depression: A systematic review of maternal and infant outcomes. Womens Health (Lond). 2019 Jan-Dec;15:1745506519844044. doi: 10.1177/1745506519844044. PMID 31035856
- [Background] Hane AA, Fox NA. Ordinary variations in maternal caregiving influence human infants' stress reactivity. Psychol Sci. 2006 Jun;17(6):550-6. doi: 10.1111/j.1467-9280.2006.01742.x. PMID 16771807
- [Background] Gunnar M, Quevedo K. The neurobiology of stress and development. Annu Rev Psychol. 2007;58:145-73. doi: 10.1146/annurev.psych.58.110405.085605. PMID 16903808
- [Background] Fan X, Wu N, Tu Y, Zang T, Bai J, Peng G, Liu Y. Perinatal depression and infant and toddler neurodevelopment: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2024 Apr;159:105579. doi: 10.1016/j.neubiorev.2024.105579. Epub 2024 Feb 10. PMID 38342472
- [Background] Kent-Marvick J, Simonsen S, Pentecost R, Taylor E, McFarland MM. Loneliness in pregnant and postpartum people and parents of children aged 5 years or younger: a scoping review. Syst Rev. 2022 Sep 7;11(1):196. doi: 10.1186/s13643-022-02065-5. PMID 36071448
- [Background] Holt-Lunstad J, Robles TF, Sbarra DA. Advancing social connection as a public health priority in the United States. Am Psychol. 2017 Sep;72(6):517-530. doi: 10.1037/amp0000103. PMID 28880099
- [Background] Mandai M, Kaso M, Takahashi Y, Nakayama T. Loneliness among mothers raising children under the age of 3 years and predictors with special reference to the use of SNS: a community-based cross-sectional study. BMC Womens Health. 2018 Aug 16;18(1):131. doi: 10.1186/s12905-018-0625-x. PMID 30111371
- [Background] Adlington K, Vasquez C, Pearce E, Wilson CA, Nowland R, Taylor BL, Spring S, Johnson S. 'Just snap out of it' - the experience of loneliness in women with perinatal depression: a Meta-synthesis of qualitative studies. BMC Psychiatry. 2023 Feb 28;23(1):110. doi: 10.1186/s12888-023-04532-2. PMID 36849948
- [Background] Wenhold H, Couture Bue AC, Kirkpatrick CE. #Bopo or Bounce Back?: Investigating the Impact of Social Media Videos on Postpartum Mothers. Health Commun. 2025 Nov;40(12):2674-2685. doi: 10.1080/10410236.2025.2475856. Epub 2025 Mar 21. PMID 40114468
- [Background] Passarelli E, Siddique M, Fry L, Hickman L, Propst K. Perineal lacerations and social media: can patients find reliable information on Instagram and TikTok? Int Urogynecol J. 2024 Jan;35(1):183-188. doi: 10.1007/s00192-023-05690-3. Epub 2023 Nov 30. PMID 38032377
- [Background] Hickman LC, Propst K, Swenson CW, Lewicky-Gaupp C. Subspecialty care for peripartum pelvic floor disorders. Am J Obstet Gynecol. 2020 Nov;223(5):709-714. doi: 10.1016/j.ajog.2020.08.015. Epub 2020 Sep 2. PMID 32888923
- [Background] McKinney J, Keyser L, Clinton S, Pagliano C. ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 Sep;132(3):784-785. doi: 10.1097/AOG.0000000000002849. No abstract available. PMID 30134408
- [Background] Priddis H, Dahlen H, Schmied V. Women's experiences following severe perineal trauma: a meta-ethnographic synthesis. J Adv Nurs. 2013 Apr;69(4):748-59. doi: 10.1111/jan.12005. Epub 2012 Oct 12. PMID 23057716
- [Background] Priddis HS, Schmied V, Kettle C, Sneddon A, Dahlen HG. "A patchwork of services"--caring for women who sustain severe perineal trauma in New South Wales--from the perspective of women and midwives. BMC Pregnancy Childbirth. 2014 Jul 18;14:236. doi: 10.1186/1471-2393-14-236. PMID 25034120
- [Background] Nutaitis AC, Ferrando CA, Propst K. Patient Perspectives Following Obstetric Anal Sphincter Injury. Urogynecology (Phila). 2025 Feb 1;31(2):161-169. doi: 10.1097/SPV.0000000000001506. Epub 2024 Apr 10. PMID 38621419
- [Background] Wallwiener S, Muller M, Doster A, Laserer W, Reck C, Pauluschke-Frohlich J, Brucker SY, Wallwiener CW, Wallwiener M. Pregnancy eHealth and mHealth: user proportions and characteristics of pregnant women using Web-based information sources-a cross-sectional study. Arch Gynecol Obstet. 2016 Nov;294(5):937-944. doi: 10.1007/s00404-016-4093-y. Epub 2016 Apr 15. PMID 27084763
- [Background] Declercq ER, Sakala C, Corry MP, Applebaum S, Herrlich A. Major Survey Findings of Listening to Mothers(SM) III: New Mothers Speak Out: Report of National Surveys of Women's Childbearing ExperiencesConducted October-December 2012 and January-April 2013. J Perinat Educ. 2014 Winter;23(1):17-24. doi: 10.1891/1058-1243.23.1.17. PMID 24453464
- [Background] Tully KP, Stuebe AM, Verbiest SB. The fourth trimester: a critical transition period with unmet maternal health needs. Am J Obstet Gynecol. 2017 Jul;217(1):37-41. doi: 10.1016/j.ajog.2017.03.032. Epub 2017 Apr 5. PMID 28390671
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Harrison V, Moore D, Lazard L. Supporting perinatal anxiety in the digital age; a qualitative exploration of stressors and support strategies. BMC Pregnancy Childbirth. 2020 Jun 17;20(1):363. doi: 10.1186/s12884-020-02990-0. PMID 32546131
- [Background] Gonzalez-Timoneda A, Valles-Murcia N, Munoz Esteban P, Torres Lopez MS, Turrion Martinez E, Errandonea Garcia P, Serrano Raya L, Nohales Alfonso F. Prevalence and impact of pelvic floor dysfunctions on quality of life in women 5-10 years after their first vaginal or caesarian delivery. Heliyon. 2025 Jan 21;11(3):e42018. doi: 10.1016/j.heliyon.2025.e42018. eCollection 2025 Feb 15. PMID 39916837
- [Background] Cassado J, Simo M, Rodriguez N, Porta O, Huguet E, Mora I, Girvent M, Fernandez R, Gich I. Prevalence of levator ani avulsion in a multicenter study (PAMELA study). Arch Gynecol Obstet. 2020 Jul;302(1):273-280. doi: 10.1007/s00404-020-05585-4. Epub 2020 May 24. PMID 32449062
- [Background] DeLancey JOL, Masteling M, Pipitone F, LaCross J, Mastrovito S, Ashton-Miller JA. Pelvic floor injury during vaginal birth is life-altering and preventable: what can we do about it? Am J Obstet Gynecol. 2024 Mar;230(3):279-294.e2. doi: 10.1016/j.ajog.2023.11.1253. Epub 2024 Jan 2. PMID 38168908
- [Background] Lien KC, Mooney B, DeLancey JO, Ashton-Miller JA. Levator ani muscle stretch induced by simulated vaginal birth. Obstet Gynecol. 2004 Jan;103(1):31-40. doi: 10.1097/01.AOG.0000109207.22354.65. PMID 14704241
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443